CLINICAL TRIAL: NCT01768351
Title: Direct Effect of Paricalcitol on Anemia in Chronic Kidney Disease
Brief Title: Paricalcitol Effect on Anemia in CKD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, Eleonora Riccio, MD, Federico II University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PCX1234; paranemia (Other: Federico II University of Naples)
Record Dates: First submitted 2013-01-13; First posted 2013-01-15 (Estimated); Last update posted 2014-07-30 (Estimated); Status verified 2012-11

CONDITIONS: Anemia; Chronic Kidney Disease
Keywords: anemia; chronic kidney disease; vitamin D; paricalcitol; hyperparathyroidism
MeSH Terms: conditions — Anemia; Renal Insufficiency, Chronic; Hyperparathyroidism | interventions — paricalcitol; Calcitriol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (Active Comparator): Patients receiving treatment for secondary hyperparathyroidism with calcitriol. The calcitriol dosage schedule provided for an initial dose of 0.5 mch every other day and titration was performed on the basis of the serum levels of intact PTH (iPTH) (target 150-300 pg/mL), Ca, P and Ca x P product as suggested by the US National Kidney Foundation Dialysis outcomes Quality Initiative (NKF-DOQI) and Kidney Disease: Improving Global Outcomes (KDIGO) guidelines.
  Interventions: Drug: Calcitriol
- Paricalcitol (Experimental): Patients treated by Paricalcitol for hyperparathyroidism. The paricalcitol initial dose was 1 mcg/die, and titration was performed on the basis of the serum levels of iPTH, Ca, P and Ca x P product as suggested by the NKF-DOQI and KDIGO guidelines.
  Interventions: Drug: Paricalcitol

INTERVENTIONS:
Drug: Paricalcitol — Zemplar cp 1 mcg/day per os
  Other Names: Zemplar
  Arms: Paricalcitol
Drug: Calcitriol — Rocaltrol cp 0,5 mcg every other day per os
  Other Names: Rocaltrol
  Arms: Control

SUMMARY:
Current activated Vitamin D therapies are approved for treating secondary hyperparathyroidism in chronic kidney disease (CKD), and a large body of experimental data in animals confirms the effects of Vitamin D that extend beyond mineral metabolism. Several studies show that the benefits are greater with the newer vitamin D analog paricalcitol when compared with calcitriol. A large gap exists in our knowledge between epidemiological studies in human that demonstrate improved outcomes with vitamin D use and observations in preclinical studies demonstrating the pleiotropic effects of Vitamin D. To explore the provenance of epidemiological outcomes in CKD, we conducted a pilot randomized trial to determine whether the use of paricalcitol, compared to calcitriol, leads to improvement in anemia, a marker associated with worse outcomes in chronic kidney disease, and whether this effect not only reflects the hyperparathyroidism correction, but is also dependent on the direct effects of paricalcitol on erythroid progenitor cells.

DETAILED DESCRIPTION:
To better understand the direct effects of paricalcitol on anemia in patients with chronic kidney disease (stage 3-5), we conducted a pilot trial in 60 patients who were randomly allocated equally to 2 groups to receive or not paricalcitol orally for 6 months.

ELIGIBILITY:
Inclusion criteria:

* age > 18
* written informed consent
* CKD stage 3-5 (eGFR <60 ml/min/1,73 m2)
* PTH 30-300 pg/ml
* Hb <10 g/dl >3 consecutive months
* Ferritin > 100 ng/ml
* transferrin saturation (TSAT) 20-40%
* mean corpuscular volume (MCV) 85-95%
* for patients treated with Ace-inhibitors or angiotensin receptor blockers, dose stable >3 months
* for patients treated with erythropoiesis-stimulating agents (ESA), dose stable >3 months

Exclusion criteria:

* anemia due to non renal cause
* presence of malignancies, inflammatory or infectious disease >3 months
* pregnancy
* bleeding >6 months
* C-reactive protein (CRP) >1 mg/dl
* poorly controlled hypertension (PAS > 170 mmHG and PAD >100 mmHg)
* severe malnutrition
* hypercalcemia (>10,5 mg/dl)
* hyperphosphatemia (>5,5 mg/dl)
* surgical interventions >3 months
* acute myocardial infarction, unstable angina, stroke or transitory ischemic attack, deep venous or pulmonary thromboembolism, congestive heart failure >3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2010-10; Primary Completion 2011-03 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Modification in hemoglobin levels | 6 months

SECONDARY OUTCOMES:
Modifications in urinary protein excretion | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Eleonora Riccio, MD, Principal Investigator
Locations (1):
- Federico II University, Naples, Italy

REFERENCES:
- [Derived] Riccio E, Sabbatini M, Bruzzese D, Capuano I, Migliaccio S, Andreucci M, Pisani A. Effect of paricalcitol vs calcitriol on hemoglobin levels in chronic kidney disease patients: a randomized trial. PLoS One. 2015 Mar 17;10(3):e0118174. doi: 10.1371/journal.pone.0118174. eCollection 2015. PMID 25781618